CLINICAL TRIAL: NCT03717961
Title: Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Study to Assess Efficacy of Botulinum Toxin A in Adult Subjects With Raynaud Phenomenon Secondary to Systemic Sclerosis
Brief Title: Efficacy of Botulinum Toxin A in Adult Subjects With Raynaud Phenomenon Secondary to Systemic Sclerosis
Acronym: BRASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P170904J
Record Dates: First submitted 2018-10-15; First posted 2018-10-24 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Raynaud Phenomenon Secondary to Systemic Sclerosis
Keywords: Raynaud Phenomenon; Systemic Sclerosis; Botulinum toxin A
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, placebo-controlled, parallel groups, phase III
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: this study is double blind masking: Both participants and investigators are unaware of the intervention assignment, others including statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- " BTX-A" group (Experimental): * BOTOX® solution
  * Saline serum
  * lidocaine/prilocaine cream
  * Nitrous oxide/oxygen (50%/50%)
  Intervention Description :
  * BOTOX 100 UNITES (Allergan, Courbevoie, France, and São Paulo, Brazil) Single injection schedule of BOTOX® in both hands, diluted in 2 ml of sterile serum saline, with a dosage of 50 UI (1 ml) by hand. Injections will be performed at the level of the distal palmar crease, targeting the neurovascular bundles in the 4 web spaces (0.25 ml/injection site)
  * between 2 to 3 hours before the procedure, application of lidocaine/prilocaine cream under an occlusive dressing (polyurethane film) in each palmar crease of the patients (1/2 tube/hand), according to the recommendations of the manufacturer
  * inhaled nitrous oxide/oxygen (50% / 50%) may be used, if needed
  Interventions: Drug: BOTOX® solution
- Placebo group (Placebo Comparator): * Saline serum
  * lidocaine/prilocaine cream
  * Nitrous oxide/oxygen (50%/50%)
  Intervention Description :
  * Sterile saline solution Single injection schedule of 2 ml (1 ml by hand) of serum saline, in both hands. Injections will be performed at the level of the distal palmar crease, targeting the neurovascular bundles in the 4 web spaces (0.25 ml/injection site).
  * between 2 to 3 hours before the procedure, application of lidocaine/prilocaine cream under an occlusive dressing (polyurethane film) in each palmar crease of the patients (1/2 tube/hand), according to the recommendations of the manufacturer of the lidocaine cream.
  * inhaled nitrous oxide/oxygen (50% / 50%) may be used, if needed
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: BOTOX® solution — Botox solution + Saline serum + lidocaine/prilocaine cream + Nitrous oxide/oxygen (50%/50%)
  Arms: " BTX-A" group
Drug: Placebo group — Placebo + lidocaine/prilocaine cream + Nitrous oxide/oxygen (50%/50%)
  Arms: Placebo group

SUMMARY:
This study aims to assess whether or not a single injection schedule of botulinum toxin A (BTX-A) in both hands improves Raynaud phenomenon (RP) secondary to systemic sclerosis (SSc) better than a placebo at 4, 12 and 24 weeks after the treatment.

This study's hypothesis is that the number of RP attacks per week from baseline to 4 weeks after treatment is significantly lower in the group treated with BTX-A than in the control group treated by the placebo. Furthermore, BTX-A in both hands is expected to improve both symptomatic (attack frequency, digital ulcer healing) and functional (pain, hand function, quality of life) symptoms of RP secondary to SSc more than placebo.

DETAILED DESCRIPTION:
In SSc, RP is present in 95% of the patients. Despite cold avoidance, RP attacks are severe, painful, affecting the quality of life, with frequent severe ischemic symptoms such as digital ulcers. Treating patients with RP secondary to SSc is extremely challenging. Oral calcium channel blockers, the most commonly prescribed drugs, were shown to be minimally effective in reducing frequency and severity of RP attacks. There is limited evidence for the efficacy of alpha-1-adrenergic receptor antagonists, angiotensin receptor blockers, phosphodiesterase inhibitors and endothelin-1 receptor antagonists to treat RP. The intravenously administered prostacyclin analogue iloprost is considered a second-line therapy, after oral calcium channel blockers, but its administration requires a 5-days hospitalisation for progressive increase in dosage and close blood pressure monitoring. Side effects are almost constant: headache, flushing, malaise and hypotension. Between 2004 and 2015, a total of 145 patients underwent botulinum toxin-A (BTX-A) injections to treat RP in case reports, retrospective or open studies. Since 2016, only 1 randomized, controlled study was performed, including 40 patients but was underpowered, not designed for clinical outcomes, and treated the patient only in one hand. Symptomatic patients treated by BTX-A experienced, in the 3 to 6 following months, pain relief in 75-100% of the cases, as well as reduction in severity and frequency of attacks and increased ulcer healing rate, with minimal adverse effects. The most common complication was temporary hand weakness, related to the injected dose. When the total dose/hand was 50 UI or lower, the rate of hand weakness was 0 to 9%. The proposed study is the first randomized double blinded multicenter clinical trial designed to assess whether or not a single injection schedule of BTX-A in both hands improves RP secondary to SSc better than a placebo at 4, 12 and 24 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Diagnosed with systemic sclerosis (EULAR/ACR 2013 criteria ; or Leroy and Metsger criteria).
* Symptoms of Raynaud's phenomenon affecting both hands (not necessarily to equal extents)
* Frequency of Raynaud's attacks ≥ 5/week during cold weather
* Stable dose of phosphodiesterase inhibitors (sildenafil, tadalafil or vardenafil), endothelin antagonists, or calcium channel blockers defined as 1-month with no change in dose
* Ability to return/be available for follow-up evaluations
* Ability to fill the diary
* Ability/willingness to give informed consent
* Affiliation to any French social security regime

Exclusion Criteria:

* History of myasthenia gravis or Eaton Lambert syndrome
* Inflammatory myositis <2 years or pre-existing motor neurone disease or upper limb motor neuropathy
* Reported allergy or hypersensitivity to any Botulinum toxin preparation or to lidocaine or other local anesthetic agent or to albumin or to inhaled nitrous oxide/oxygen.
* Active infection in either hand.
* Pregnant or lactating women (women of child bearing potential must undergo a urine pregnancy teste before inclusion and at treatment day).
* women of child bearing potential without medically accepted method of birth control
* Patients who have previously undergone any vascular surgery on the upper extremity, including surgical sympathectomy or ever received botulinum toxin or planned to receive botulinum toxin in the next 6 months
* Cognitive impairment
* Iloprost scheduled the month following injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in the number of RP attacks per week at 4 weeks | 4 weeks
  Comparison between the 2 groups of the change (absolute) from baseline in the number of RP attacks per week at 4 weeks. An attack is defined as an episode of pallor or cyanosis (with or without pain, tingling or numbness). Subjects will keep a daily record of the number of RP attacks they experienced per day and the duration of each attack, from Day -14 to Day 0 (+/- 4 days) and from Day 14 to Day 28 ( +/- 4 days)

SECONDARY OUTCOMES:
Absolute change from baseline in the number of RP attacks per week at 12 and 24 weeks | 24 weeks
  Comparison between the 2 groups of the change (absolute) from baseline in the number of RP attacks per week at 12 and 24 weeks. Subjects kept a daily record of the number of RP attacks they experienced per day and the duration of each attack, over a 14-day +/- 4 days period before each assessment visit at 12 and 24 weeks
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the percentage of digital ulcers with complete healing | 24 weeks
  Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the percentage of digital ulcers with complete healing
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the number of new digital ulcers. | 24 weeks
  Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the number of new digital ulcers.
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in Raynaud's pain score. | 24 weeks
  Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in Raynaud's pain score. Pain associated with each attack is self-reported on a 10-point scale, and averaged over 14-day +/- 4 days period before each assessment visit
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in Raynaud's Condition Score. | 24 weeks
  Comparison at 4, 12 and 24 weeks of follow-up after the treatment of the change in Raynaud's Condition Score. Raynaud Condition Score is a daily self-assessment of RP activity using a 0-10 ordinal scale and averaged over 14-day +/- 4 days period before each assessment visit. The RCS incorporates the cumulative daily frequency, duration, severity and impact of RP attacks.
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in quality of life from baseline to weeks 4, 12 and 24 | 24 weeks
  Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in quality of life from baseline to weeks 4, 12 and 24. QOL is assessed by the Health Assessment Questionnaire (HAQ)
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in hand function from baseline to weeks 4, 12 and 24 | 24 weeks
  Comparison between the 2 groups from baseline to 4, 12 and 24 weeks of follow-up after the treatment of the change in hand function measured by Quick-DASH (Disabilities of the Arm, Shoulder and Hand)
Comparison between the 2 groups at 4, 12 and 24 weeks of follow-up after the treatment of the change in hand function from baseline to weeks 4, 12 and 24 | 24 weeks
  Comparison between the 2 groups from baseline to at 4, 12 and 24 weeks of follow-up after the treatment of the change in hand function measured by the Hand Function Scale of Cochin
Frequency and severity of adverse drug events during treatment from baseline to weeks 4, 12 and 24. | 24 weeks
  Frequency and severity of adverse drug events during treatment from baseline to weeks 4, 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Senet, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Senet P, Maillard H, Diot E, Lazareth I, Blaise S, Arnault JP, Pistorius MA, Boulon C, Cogrel O, Warzocha U, Riviere S, Malloizel-Delaunay J, Servettaz A, Sassolas B, Viguier M, Monfort JB, Janique S, Vicaut E; BRASS collaborators. Efficacy and Safety of Botulinum Toxin in Adults with Raynaud's Phenomenon Secondary to Systemic Sclerosis: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study. Arthritis Rheumatol. 2023 Mar;75(3):459-467. doi: 10.1002/art.42342. Epub 2022 Dec 14. PMID 36066501